CLINICAL TRIAL: NCT03295305
Title: Effect of Action-Based Cognitive Remediation on Cognition and Frontal Lobe Activity in Patients With Bipolar Disorder in Remission (PRETEC-ABC)
Brief Title: Effect of Action-Based Cognitive Remediation in Patients With Bipolar Disorder
Acronym: PRETEC-ABC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Collaborators: Lundbeck Foundation (Other)
Responsible Party: Principal Investigator, Kamilla Woznica Miskowiak, Professor, Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-16043480; 2012-58-0004 (Registry Identifier: Danish Data Protection Agency)
Record Dates: First submitted 2017-09-15; First posted 2017-09-27 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Bipolar Disorder; Cognitive Impairment
Keywords: Biomarker; Bipolar Disorder; Cognition; Cognitive Impairment; cognitive remediation; functional magnetic resonance imaging; pro-cognitive effect
MeSH Terms: conditions — Bipolar Disorder; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Action Based Cognitive Remediation (Experimental)
  Interventions: Behavioral: Action-Based Cognitive Remediation
- Unstructured support group (Active Comparator)
  Interventions: Behavioral: Unstructured support group

INTERVENTIONS:
Behavioral: Action-Based Cognitive Remediation
  Arms: Action Based Cognitive Remediation
Behavioral: Unstructured support group
  Arms: Unstructured support group

SUMMARY:
PRETEC-ABC aims to assess the effect of a new form of cognitive remediation, Action-Based Cognitive Remediation (ABCR), in patients with bipolar disorder in remission on cognition, and to assess the neural assays for treatment effects with the purpose of identifying a neural biomarker for pro-cognitive effect. It is hypothesized (i) that ABCR vs. a control treatment has a beneficial effect on cognition in remitted patients with bipolar disorder remission. It is hypothesized (ii) that this treatment-associated improvement of cognition translates into better functional capacity at a six months follow-up assessment (secondary outcome). Finally, as an exploratory measure, it is hypothesized that ABCR will produce an early change in frontal activity and that this activity will correlate with ABCR-associated improvements in cognitive function.

DETAILED DESCRIPTION:
The trial will include outpatients with BD in full or partial remission (a score ≤14 on the Hamilton Depression Rating Scale (HDRS) and Young Mania Rating Scale (YMRS). Recruitment will be carried out through the ongoing Bipolar Illness Onset (BIO) study, the Copenhagen Affective Disorder Clinic, Psychiatric Centre Copenhagen, Rigshospitalet, other mental health centres, consultant psychiatrists in the Capital Region of Denmark, and through advertisements on relevant websites.

Participants will undergo an eligibility assessment followed by randomisation. When 4 - 6 participants have been randomised to either the ABCR or the control group, the baseline assessments are carried out. The baseline assessment is completed over two days, 1 - 3 days apart. A fMRI scan is carried out on day 1 encompassing spatial and verbal working memory N-back tasks, a picture encoding task, a resting state and a structural scan. On day 2, a blood sample is drawn in the morning, followed by administration of a comprehensive neuropsychological test battery. Participants fill in questionnaires concerning subjective cognitive complaints, psychosocial functioning and quality of life and functional capacity is assessed using a clinician-rated interview and a performance based assessment. Sleep quantity and quality in the past three days is assessed. After two weeks of ABCR or control treatment, functional MRI, neuropsychological testing an assessment of mood and subjective cognition are repeated. These assessments, as well as assessments of functional capacity and quality of life, are repeated within two weeks after treatment completion and six months after treatment completion.

Block randomisation is carried out by Pharma Consulting Group, stratified by gender and age (patients < or ≥ 35 years).

Power calculation was also carried out by Pharma Consulting Group based on findings from a previous RCT in our group assessing the effect of 8 weeks of EPO treatment on the same cognitive composite score. In PreTEC-ABC, a clinically relevant difference between the ABCR and the control groups following 10 weeks of treatment is assumed to be 0.4 SD (corresponding to a medium effect size) on the primary outcome, with a mean change in the cognitive composite score of 0.5 SD. Assuming a 10% drop-out rate, we will recruit up to N=58 in order to achieve complete datasets for N=52 participants.

Data will be analysed using mixed models using intention-to-treat (ITT) analyses.

Functional MRI-data will be pre-processed and analysed with the FMRIB Expert Analysis Tool (FEAT) and the "randomize" algorithm implemented in FMRIB Software Library (FSL). Functional MRI data will be analysed using a Region of interest (ROI) analysis to assess differences between the ABCR and control group in neural activity in the dlPFC and the hippocampi after 2 weeks. Exploratory whole-brain analyses will be conducted to investigate any effects in other brain regions. Any differences in neural activity will be correlated with potential changes in the cognitive composite score at weeks 2 and post-treatment. If there is a significant correlation with cognition at post-treatment, multiple regression analysis will be carried out, adjusting for mood and demographic characteristics, to assess whether early change in neural activity is predictive of pro-cognitive effects.

ELIGIBILITY:
Inclusion Criteria:

* Fluent Danish skills and objective cognitive impairment (a total score below cutoff, or scores below cutoff on a minimum of two out of the five subtests (Verbal Learning Test - Immediate, Working Memory Test, Verbal Fluency Test, Verbal Learning Test - Delayed and Processing Speed Test) on the Screen for Cognitive Impairment in Psychiatry - Danish version (SCIP-D).
* Patients must meet the ICD-10 diagnosis of BD (type I and II) confirmed using the Schedules for Clinical Assessment in Neuropsychiatry (SCAN) interview.

Exclusion Criteria:

* Daily use of benzodiazepines > 22.5 mg oxazepam, pregnancy, current drug or substance abuse (three months prior to inclusion), previous serious head trauma, severe physical illness, neurological illness, schizophrenia or schizoaffective disorder, dyslexia, claustrophobia, having a pacemaker or other metal implants inside the body and electroconvulsive therapy in the three months prior to inclusion.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2020-01-25 (Actual)

PRIMARY OUTCOMES:
Cognitive composite score | Change from baseline and week 11
  A cognitive composite based on an average of the Rey Auditory Verbal Learning Test (RAVLT), Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) Coding, verbal fluency with the letter "D", WAIS-III Letter-Number Sequencing, Trail Making Test B (TMT B) and Rapid Visual Information Processing (RVP) from Cambridge Cognition (CANTAB).

SECONDARY OUTCOMES:
One Touch Stockings of Cambridge | Baseline, two weeks of treatment, week 11, and 6-months follow-up
  A computerized neuropsychological test assessing executive functions
Functional Assessment Short Test | Baseline, week 11, and 6-months follow-up
  A semi-structured interview assessing level of functioning

OTHER OUTCOMES:
Rey Auditory Verbal Learning Test | Baseline, two weeks of treatment, week 11, and 6-months follow-up
  Neuropsychological test assessing verbal memory
Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) Coding | Baseline, two weeks of treatment, week 11, and 6-months follow-up
  Neuropsychological test assessing attention
Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) Digit Span | Baseline, two weeks of treatment, week 11, and 6-months follow-up
  Neuropsychological test assessing executive functions
Verbal fluency with the letter "D" and 'S" | Baseline, two weeks of treatment, week 11, and 6-months follow-up
  Neuropsychological test assessing executive functions
WAIS-III Letter-Number Sequencing | Baseline, two weeks of treatment, week 11, and 6-months follow-up
  Neuropsychological test assessing executive functions
Trail Making Test B | Baseline, two weeks of treatment, week 11, and 6-months follow-up
  Neuropsychological test assessing psychomotor speed
Trail Making Test A | Baseline, two weeks of treatment, week 11, and 6-months follow-up
  Neuropsychological test assessing executive functions
Rapid Visual Information Processing (RVP) from Cambridge Cognition (CANTAB) | Baseline, two weeks of treatment, week 11, and 6-months follow-up
  Neuropsychological test assessing sustained attention
Spatial Working Memory (SWM) from Cambridge Cognition | Baseline, two weeks of treatment, week 11, and 6-months follow-up
  Neuropsychological test assessing sustained attention
Brief University of California, San Diego Performance-Based Skills Assessment-B (UPSA-B) | Baseline, week 11, and 6-months follow-up
  Objective assessment of level of functioning
Sheehan Disability Scale | Baseline, week 11, and 6-months follow-up
  Questionnaire on level of functioning
The Assessment of Quality of Life | Baseline, week 11, and 6-months follow-up
  Questionnaire on quality of life
World Health Organization Quality of Life (WHOQOL-BREF) | Baseline, week 11, and 6-months follow-up
  Questionnaire on quality of life
Cognitive Complaints in Bipolar Disorder Rating Assessment (COBRA) | Baseline, two weeks of treatment, week 11,and 6-months follow-up
  Questionnaire on subjective cognitive complaints
Work and Social Adjustment Scale (WSAS) | Baseline, week 11, and 6-months follow-up
  Questionnaire on occupational functioning

CONTACTS AND LOCATIONS:
Overall Officials: Kamilla W Miskowiak, Dr, Principal Investigator — Mental Health Services, Capital Region of Denmark
Locations (1):
- Mental Health Services, Capital Region of Denmark, Copenhagen University Hospital, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ott CV, Vinberg M, Kessing LV, Bowie CR, Forman JL, Miskowiak KW. Effect of Action-Based Cognitive Remediation on cognitive impairment in patients with remitted bipolar disorder: A randomized controlled trial. Bipolar Disord. 2021 Aug;23(5):487-499. doi: 10.1111/bdi.13021. Epub 2020 Oct 29. PMID 33053258
- [Derived] Ott CV, Vinberg M, Bowie CR, Christensen EM, Knudsen GM, Kessing LV, Miskowiak KW. Effect of action-based cognitive remediation on cognition and neural activity in bipolar disorder: study protocol for a randomized controlled trial. Trials. 2018 Sep 12;19(1):487. doi: 10.1186/s13063-018-2860-8. PMID 30208971